CLINICAL TRIAL: NCT03013153
Title: Low or High Ligation of the Inferior Mesenteric Artery With Apical Lymph Node Dissection in Rectal Cancer Laparoscopic Surgery: A Prospective, Multi-Center, Randomized, Open-Label, Parallel Group, Non-Inferiority Clinical Trial (LAND)
Brief Title: Low or High Ligation of the IMA With Apical Lymph Node Dissection in Rectal Cancer Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAND
Record Dates: First submitted 2016-12-31; First posted 2017-01-06 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-12

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Inferior Mesenteric Artery; Ligation; Apical Lymph Nodes; Laparoscopy; IMA Types
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low ligation with apical lymph node dissection (Experimental): Left colic artery (LCA) is identified according to the CT 3D-reconstruction, tie the sigmoid artery and superior rectal artery, preserved LCA while low ligation of the inferior mesenteric artery is performed. Lymphadenectomy to the apical lymph nodes (No.253)is performed around the IMA until 2 cm from the aorta. The inferior mesenteric vein (IMV) is divided and ligated below the pancreatic margin.
  Interventions: Procedure: Low ligation with apical lymph node dissection
- High ligation (Active Comparator): Open the peritoneum proceeds cephalad towards the duodenojejunal angle of Treitz, and the mesenteric root is incised 1 cm below the inferior margin of the pancreas. The aortomesenteric window is opened wide and the inferior mesenteric vessels are exposed. The IMA is ligated and divided at 2 cm from its origin. The inferior mesenteric vein (IMV) is divided and ligated below the pancreatic margin.
  Interventions: Procedure: High ligation

INTERVENTIONS:
Procedure: Low ligation with apical lymph node dissection — Low ligation with apical lymph node dissection (LAND). Left colic artery (LCA) is identified according to the CT 3D-reconstruction, tie the sigmoid artery and superior rectal artery, preserved LCA while low ligation of the inferior mesenteric artery is performed. Lymphadenectomy to the apical lymph nodes (No.253)is performed around the IMA until 2 cm from the aorta.
  Other Names: LAND
  Arms: Low ligation with apical lymph node dissection
Procedure: High ligation — High ligation (HL) Open the peritoneum proceeds cephalad towards the duodenojejunal angle of Treitz, and the mesenteric root is incised 1 cm below the inferior margin of the pancreas. The aortomesenteric window is opened wide and the inferior mesenteric vessels are exposed. The IMA is ligated and divided at 2 cm from its origin. The inferior mesenteric vein (IMV) is divided and ligated below the pancreatic margin.
  Other Names: HL
  Arms: High ligation

SUMMARY:
Laparoscopy colon surgery is accepted worldwide in the recent years. But there is still argument on the effect of laparoscopy rectal surgery. Laparoscopy has advantages on showing the inferior mesenteric artery (IMA), protection of autonomic nerve, low rectal anastomosis, and total mesorectum excision. However, debate on the level of IMA ligation and debonding of splenic flexure never ends. This study is going to give a clear and definite answer to how and why surgeons should deal with the IMA in laparoscopy rectal surgery，base on the 3D reconstruction of IMA and identification of IMA perfusion types.

DETAILED DESCRIPTION:
According to the report of World Health Organization 2015, the morbility and mortality of colorectal cancer (CRC) are rising all over the world. Although the technique gets great approval in CRC surgical treatment in the recent years, such as TME protocol, neoadjuvant and laparoscopy technique, the complication of anastomosis leakage and nerve damage are still to be solved.

Laparoscopy colon surgery is accepted worldwide in the recent years. But there is still argument on the effect of laparoscopy rectal surgery. Laparoscopy has advantages on showing the inferior mesenteric artery, protection of autonomic nerve, low rectal anastomosis, and total mesorectum excision. However, debate on where is the best level of IMA ligation and whether splenic flexure be debonded never ends. This study is going to give a clear and definite answer to how and why surgeons should deal with the IMA in laparoscopy rectal surgery.

The ligation level of IMA affects on hypogastric and pelvic nerve, leads to disorder of sexual and urination functions. What's more, it also have affection on the apical lymph node (No.253) harvesting and the blood supplement of proximal colon. Former studies have proved that the blood supplement and tension of anastomosis leads to leakage after surgery. Meanwhile, the ligation level of IMA is the key point on it.

The former study comes from the sixth affiliated hospital found that the mistake of ligation level of IMA happened because of the poor touching and explosion with laparoscopy. The distance from the root of IMA to left colic artery (DRL) vary between 19mm and 64mm. When surgeon made mistake during ligation, it led to the insufficient resection of apical lymph node. Further more, affect the long-term survival. Besides, there are 4 different types of IMA according to the relationship between the left colic artery, sigmoid artery and superior rectal artery. These branches will confuse surgeon on how to deal with them. 3D reconstruction of abdominal pelvic CT is able to show the length of DRL, IMA types and apical lymph nodes clearly. With these technique, the investigators can preserve the left colic artery and resect apical lymph nodes precisely.

In the past studies, high or low ligation takes advantage on both side. But none of them comes from retrospective clinical trail. Some author believe that high ligation do better in resection of apical lymph nodes, release the tension of anastomosis, providing precise tumor staging. On the other side, some authors consider that high ligation may cut down blood supplement, rise the incident of anastomosis leakage (AL). so they prefer low ligation to the high. Some studies show that there are no long term survival difference between high and low ligation on IMA in laparoscopy rectal resection. So whether high ligation is necessary, still to be proved.

For local advanced rectal cancer, neoadjuvant chemotherapy can lesson tumor size, reduce recurrence, preserve annual better and rise long-term survival. National Comprehensive Cancer Network command chemotherapy before surgery (Total Mesorectal Excision TME) as the standard for rectal cancer since 2005. Another randomized controlled trial (RCT) named Neoadjuvant FOLFOX6 Chemotherapy With or Without Radiation in Rectal Cancer (FOWARC) NCT01211210 has proved the recent positive result. In those cases, the positive metastasis apical lymph node appeared in less than 5% (5/116) cases. On the other side, the incident of AL was up to 7% (8/116) . This phenomenon discover that maybe low ligation with apical lymph nodes dissection can get the same treatment effect and decrease AL from happening.

ELIGIBILITY:
Inclusion Criteria:

* Pathology shows rectal or sigmoid adenocarcinoma
* The bottom edge of tumor to anuas is less than 15cm
* The clinical staging of tumor by American Joint Committee on Cancer (AJCC) within T2-4 or N1-2
* Receive or not receive neoadjuvant chemotherapy based on 5-fluorouracil before surgery
* Racial resection in available after neoadjuvant chemotherapy
* No metastasis evidence was found
* Annual preservation surgery is available
* Tolerate to general anesthesia
* Eastern Cooperative Oncology Group (ECOG) status score between 0 and 1
* Patients and general anesthesia can understand the clinical trail well and are willing to take part in

Exclusion Criteria:

* Suffer with other carcinoma synchronous or metachronous in 5 years
* Multiple primary colon carcinoma
* Radiation therapy was performed before surgery
* History of colorectal surgery
* Combine with acute intestinal obstruction, intestinal bleeding, intestinal perforation and emergency surgery is needed
* Multiple organs resection surgery is needed
* Abdominal perineal resection is performed
* American Society of Anesthesiologists score stage IV to V
* Pregnant, suckling period or reject to contraception
* Severe cardiovascular disease, uncontrollable infection or other severe complication
* Severe mental illness
* Unable to go through the treatment because of family, society or regional condition
* Refuse to take part in the trail

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
5-years overall survival rate | 5 years
  5-years overall survival rate

SECONDARY OUTCOMES:
5-years disease free survival rate | 5 years
  5-years disease free survival rate
1-year overall survival rate | 1 year
  1-year overall survival rate
1-year disease free survival rate | 1 year
  1-year disease free survival rate
Anastomosis leakage rate | 6 months
  anastomosis leakage rate after surgery, acute or chronic
Apical Lymph Nodes (LN) Positive Rate | 1 week
  Apical Lymph Nodes Positive Rate, No.253 LN
Operation Time | 1 day
Blood loss during operation | 1 day
Complication incident rate of surgery | 1 day
conversion rate to laparotomy | 1 day
Identification of IMA perfusion type before surgery | 1 day
Identification of lymph node metastasis by CT | 7 days
Mortality rate in 30 days after surgery | 30 days
Recovery time after surgery | 60 days
White cell level | 7 days
C-reaction protein level | 7 days
Albumin level | 7 days
Anastomosis bleeding rate after surgery | 30 days
Anastomosis stenosis rate after surgery | 30 days
Intestinal dysfunction after stoma closure | 1 year
Anus function after surgery | 1 year
Life quality scoring | 1 year
Bladder residual urine volume | 1 year
Sexual function scoring | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Meijin Huang, MD, Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The sixth affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mari G, Maggioni D, Costanzi A, Miranda A, Rigamonti L, Crippa J, Magistro C, Di Lernia S, Forgione A, Carnevali P, Nichelatti M, Carzaniga P, Valenti F, Rovagnati M, Berselli M, Cocozza E, Livraghi L, Origi M, Scandroglio I, Roscio F, De Luca A, Ferrari G, Pugliese R. "High or low Inferior Mesenteric Artery ligation in Laparoscopic low Anterior Resection: study protocol for a randomized controlled trial" (HIGHLOW trial). Trials. 2015 Jan 27;16:21. doi: 10.1186/s13063-014-0537-5. PMID 25623323
- [Background] Bostrom P, Haapamaki MM, Matthiessen P, Ljung R, Rutegard J, Rutegard M. High arterial ligation and risk of anastomotic leakage in anterior resection for rectal cancer in patients with increased cardiovascular risk. Colorectal Dis. 2015 Nov;17(11):1018-27. doi: 10.1111/codi.12971. PMID 25851151
- [Background] Tanaka J, Nishikawa T, Tanaka T, Kiyomatsu T, Hata K, Kawai K, Kazama S, Nozawa H, Yamaguchi H, Ishihara S, Sunami E, Kitayama J, Watanabe T. Analysis of anastomotic leakage after rectal surgery: A case-control study. Ann Med Surg (Lond). 2015 May 11;4(2):183-6. doi: 10.1016/j.amsu.2015.05.002. eCollection 2015 Jun. PMID 26042185
- [Background] Dauser B, Herbst F. Diagnosis, management and outcome of early anastomotic leakage following colorectal anastomosis using a compression device: is it different? Colorectal Dis. 2014 Dec;16(12):O435-9. doi: 10.1111/codi.12742. PMID 25132419
- [Background] GRIFFITHS JD. Surgical anatomy of the blood supply of the distal colon. Ann R Coll Surg Engl. 1956 Oct;19(4):241-56. No abstract available. PMID 13363265
- [Background] Masoni L, Mari FS, Nigri G, Favi F, Gasparrini M, Dall'Oglio A, Pindozzi F, Pancaldi A, Brescia A. Preservation of the inferior mesenteric artery via laparoscopic sigmoid colectomy performed for diverticular disease: real benefit or technical challenge: a randomized controlled clinical trial. Surg Endosc. 2013 Jan;27(1):199-206. doi: 10.1007/s00464-012-2420-3. Epub 2012 Jun 26. PMID 22733197
- [Background] Hida J, Okuno K. High ligation of the inferior mesenteric artery in rectal cancer surgery. Surg Today. 2013 Jan;43(1):8-19. doi: 10.1007/s00595-012-0359-6. Epub 2012 Oct 7. PMID 23052748
- [Background] Murono K, Kawai K, Kazama S, Ishihara S, Yamaguchi H, Sunami E, Kitayama J, Watanabe T. Anatomy of the inferior mesenteric artery evaluated using 3-dimensional CT angiography. Dis Colon Rectum. 2015 Feb;58(2):214-9. doi: 10.1097/DCR.0000000000000285. PMID 25585080
- [Background] Seike K, Koda K, Saito N, Oda K, Kosugi C, Shimizu K, Miyazaki M. Laser Doppler assessment of the influence of division at the root of the inferior mesenteric artery on anastomotic blood flow in rectosigmoid cancer surgery. Int J Colorectal Dis. 2007 Jun;22(6):689-97. doi: 10.1007/s00384-006-0221-7. Epub 2006 Nov 3. PMID 17082922
- [Background] Battal B, Hamcan S, Akgun V, Bozkurt Y. Congenital superior-inferior mesenteric arterial variation or arc of Riolan due to occlusion of proximal superior mesenteric artery. Surg Radiol Anat. 2014 Apr;36(3):309-10. doi: 10.1007/s00276-013-1212-3. Epub 2013 Oct 18. No abstract available. PMID 24135762
- [Background] van Gulik TM, Schoots I. Anastomosis of Riolan revisited: the meandering mesenteric artery. Arch Surg. 2005 Dec;140(12):1225-9. doi: 10.1001/archsurg.140.12.1225. PMID 16365247
- [Background] Bertrand MM, Delmond L, Mazars R, Ripoche J, Macri F, Prudhomme M. Is low tie ligation truly reproducible in colorectal cancer surgery? Anatomical study of the inferior mesenteric artery division branches. Surg Radiol Anat. 2014 Dec;36(10):1057-62. doi: 10.1007/s00276-014-1281-y. Epub 2014 Mar 15. PMID 24633578
- [Background] Trencheva K, Morrissey KP, Wells M, Mancuso CA, Lee SW, Sonoda T, Michelassi F, Charlson ME, Milsom JW. Identifying important predictors for anastomotic leak after colon and rectal resection: prospective study on 616 patients. Ann Surg. 2013 Jan;257(1):108-13. doi: 10.1097/SLA.0b013e318262a6cd. PMID 22968068
- [Background] Hirst NA, Tiernan JP, Millner PA, Jayne DG. Systematic review of methods to predict and detect anastomotic leakage in colorectal surgery. Colorectal Dis. 2014 Feb;16(2):95-109. doi: 10.1111/codi.12411. PMID 23992097
- [Background] Silberhumer GR, Paty PB, Temple LK, Araujo RL, Denton B, Gonen M, Nash GM, Allen PJ, DeMatteo RP, Guillem J, Weiser MR, D'Angelica MI, Jarnagin WR, Wong DW, Fong Y. Simultaneous resection for rectal cancer with synchronous liver metastasis is a safe procedure. Am J Surg. 2015 Jun;209(6):935-42. doi: 10.1016/j.amjsurg.2014.09.024. Epub 2014 Dec 13. PMID 25601556
- [Background] Hadidi AT. A technique to improve vascularity in colon replacement of the esophagus. Eur J Pediatr Surg. 2006 Feb;16(1):39-44. doi: 10.1055/s-2006-923925. PMID 16544225
- [Background] Raboei EH, Luoma R. Colon patch esophagoplasty: an alternative to total esophagus replacement? Eur J Pediatr Surg. 2008 Aug;18(4):230-2. doi: 10.1055/s-2008-1038396. Epub 2008 Jul 15. PMID 18629764
- [Background] Cirocchi R, Trastulli S, Farinella E, Desiderio J, Vettoretto N, Parisi A, Boselli C, Noya G. High tie versus low tie of the inferior mesenteric artery in colorectal cancer: a RCT is needed. Surg Oncol. 2012 Sep;21(3):e111-23. doi: 10.1016/j.suronc.2012.04.004. Epub 2012 Jul 6. PMID 22770982
- [Background] Gervaz P, Platon A, Buchs NC, Rocher T, Perneger T, Poletti PA. CT scan-based modelling of anastomotic leak risk after colorectal surgery. Colorectal Dis. 2013;15(10):1295-300. doi: 10.1111/codi.12305. PMID 23710555
- [Background] Doeksen A, Tanis PJ, Wust AF, Vrouenraets BC, van Lanschot JJ, van Tets WF. Radiological evaluation of colorectal anastomoses. Int J Colorectal Dis. 2008 Sep;23(9):863-8. doi: 10.1007/s00384-008-0487-z. Epub 2008 Jun 17. PMID 18560844
- [Background] Hu X, Cheng Y. A Clinical Parameters-Based Model Predicts Anastomotic Leakage After a Laparoscopic Total Mesorectal Excision: A Large Study With Data From China. Medicine (Baltimore). 2015 Jul;94(26):e1003. doi: 10.1097/MD.0000000000001003. PMID 26131798
- [Background] Qu H, Liu Y, Bi DS. Clinical risk factors for anastomotic leakage after laparoscopic anterior resection for rectal cancer: a systematic review and meta-analysis. Surg Endosc. 2015 Dec;29(12):3608-17. doi: 10.1007/s00464-015-4117-x. Epub 2015 Mar 6. PMID 25743996
- [Background] Majbar MA, Elmalki Hadj O, Souadka A, El Alaoui M, Sabbah F, Raiss M, Hrora A, Ahallat M. Risk factors for anastomotic leakage after anterior resection for rectal adenocarcinoma. Tunis Med. 2014 Jul;92(7):493-6. PMID 25775290